CLINICAL TRIAL: NCT05402033
Title: Enhancement of Access to and Diversity in Cancer Clinical Trials Through a Financial Reimbursement and Outreach Program
Brief Title: Cancer Clinical Trials Financial Reimbursement Program
Status: Recruiting | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Cancer Prevention Research Institute of Texas (Other)
Responsible Party: Principal Investigator, David E Gerber, Professor, Internal Medicine, University of Texas Southwestern Medical Center
Other Study IDs: STU-2021-1144
Record Dates: First submitted 2022-05-24; First posted 2022-06-02 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Cancer Clinical Trials
MeSH Terms: interventions — Surveys and Questionnaires; Interviews as Topic

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Survey / Interview Group: All patients (or parent / caregiver, if relevant) who provide informed consent will be asked to complete baseline assessments utilizing validated questionnaires administered through the phone or video call. The clinical research coordinator will input responses into REDCap. Alternatively, patients may request assessments be sent through secure email.
  Baseline assessment consisting of sociodemographic items and study eligibility questions (call #1)
  In addition, each patient will complete the Comprehensive Score for financial Toxicity Patient Reported Outcome Measure (COST PROM) and Short Assessment of Health Literacy (SAHL) survey measures.
  Interventions: Behavioral: Survey / Interview Group

INTERVENTIONS:
Behavioral: Survey / Interview Group — Patients with any cancer type who are informed that they may be eligible for participation in any phase therapeutic cancer clinical trial by their treating physician (typically a clinical oncologist) will be provided information about the Financial Reimbursement Program. Patients who enroll to therapeutic cancer clinical trial will be eligible for the reimbursement program and offered an opportunity to participate in this study.

SUMMARY:
To implement a Financial Reimbursement and Outreach Program at clinical sites within the Harold C. Simmons Comprehensive Cancer Center; and evaluate the impact of the program on clinical trial enrollment and demographics, as well as facilitators of and barriers to program participation.

DETAILED DESCRIPTION:
The overall purpose of this study is to determine the impact of a Financial Reimbursement Program on recruitment and retention to therapeutic cancer clinical trials, including evaluating program facilitators and barriers, as well as patient acceptability and adoption of the program.

The procedures involved for this study are surveys and interviews. Subjects will complete two surveys which are expected to take about 10-15 minutes. Some of the subjects will also be invited to complete follow-up interviews after 21 days and between 30 and 90 days. The surveys and interviews are for research purposes only.

Statistical analysis: Two-sample t-tests and chi-square tests to determine the association between socio-demographic variables, financial toxicity, health literacy, and Financial Reimbursement Program participation.

ELIGIBILITY:
Inclusion Criteria:

* Be enrolled in a therapeutic cancer clinical trial
* Speak English or Spanish

Exclusion Criteria:

* Not enrolled in a clinical trial
* Does not speak English or Spanish

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants will be recruited from among patients seen in the cancer clinics of the Harold C. Simmons Comprehensive Cancer Center, including those at UT Southwestern Medical Center, Parkland Health and Hospital System, and Children's Health. Patients with any cancer type who are informed that they are eligible for participation in any phase therapeutic cancer clinical trial by their treating physician (generally a medical oncologist) will be offered the opportunity to determine if they are interested in and eligible for the Financial Reimbursement Program and this Research Study to evaluate the Program.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2022-07-12 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Clinical trial enrollment retention rate measured by COST PROM | Up to first 60 days after enrollment to a therapeutic cancer trial.
  Use COST PROM to calculate the clinical trial enrollment and retention rates of the patients eligible for and participate in the Financial Reimbursement Program (FRP) versus those that decline to participate in the FRP.
Clinical trial enrollment retention rate measured by SAHL | Up to first 60 days after enrollment to a therapeutic cancer trial.
  Use SAHL to calculate the clinical trial enrollment and retention rates of the patients eligible for and participate in the Financial Reimbursement Program (FRP) versus those that decline to participate in the FRP.
Sociodemographic characteristics of the patients measured by COST PROM | Up to first 60 days after enrollment to a therapeutic cancer trial.
  Use COST PROM to determine the sociodemographic characteristics of the patients eligible for and participate in the Financial Reimbursement Program (FRP) versus those that decline to participate in the FRP.
Sociodemographic characteristics of the patients measured by SAHL | Up to first 60 days after enrollment to a therapeutic cancer trial.
  Use SAHL to determine the sociodemographic characteristics of the patients eligible for and participate in the Financial Reimbursement Program (FRP) versus those that decline to participate in the FRP.
Characteristics of patients enrolled in a Financial Reimbursement Program who do versus do not submit expense documentation for reimbursement | Up to first 60 days after enrollment to a therapeutic cancer trial.
  The Financial Reimbursement Program will provide monthly de-identified reports to the Project team on reimbursed expenses by category, and total dollars reimbursed, stratified by study participation. Categories of financial needs/expenses are hotels, flights, parking, gas, tolls, travel companion, bus, subway, taxi/ride hailing app, car/boat service, childcare, internet access, and miscellaneous.
Identify impact of participation in a Financial Reimbursement Program | Up to first 60 days after enrollment to a therapeutic cancer trial.
  Use COST PROM questionnaires to determine factors affecting patient participation decisions .

CONTACTS AND LOCATIONS:
Overall Officials: David E Gerber, MD, Principal Investigator — Professor
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No